CLINICAL TRIAL: NCT02351180
Title: A Randomized Placebo Controlled Trial of Inhaled Beclomethasone After Community-acquired Respiratory Viral Infection in Lung Transplant Recipients
Brief Title: Inhaled Beclomethasone After Community-Acquired Respiratory Viral Infection in Lung Transplant Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WUIBCARV1-201404080
Record Dates: First submitted 2015-01-26; First posted 2015-01-30 (Estimated); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-01

CONDITIONS: Lung Transplant Infection
Keywords: Chronic lung allograft dysfunction; Community-acquired respiratory viral infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled beclomethasone (Experimental): Inhaled beclomethasone 320 mcg twice daily for 180 days.
  Interventions: Drug: Inhaled beclomethasone
- Placebo (Placebo Comparator): Inhaled placebo twice daily for 180 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled beclomethasone — Inhaled steroid that may decrease airway inflammation and the risk of chronic rejection
  Arms: Inhaled beclomethasone
Drug: Placebo — Placebo will serve as a control treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the use of inhaled beclomethasone after a community-acquired respiratory viral infection in a lung transplant recipient decreases the risk of the subsequent development of chronic lung allograft dysfunction.

DETAILED DESCRIPTION:
Community-acquired respiratory viral (CARV) infections after lung transplantation are associated with an increased risk for the development of chronic lung allograft dysfunction (CLAD) after lung transplantation. The exact mechanisms whereby CARV infections increase this risk are unknown. We propose that viral infection results in airway epithelial cell injury and the expression of injury-response genes that provide signals that initiate immunologic and non-immunologic pathways that result in the airway remodeling characteristic of obliterative bronchiolitis, the predominant pathology of CLAD. Systemic and inhaled corticosteroids are frequently used as anti-inflammatory agents to treat the peribronchiolar inflammation seen in viral bronchiolitis. Beneficial effects from corticosteroids have been reported, but this has not been demonstrated in lung transplant recipients. The aim of this single center, randomized, double blind, placebo controlled study is to evaluate the short and long term effects of a 6 month course of inhaled beclomethasone on adult lung transplant recipients with CARV infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old)
* Single, bilateral, or heart-lung transplant recipient
* Confirmed infection with a community-acquired respiratory virus including: adenovirus, coronavirus, influenza A or B, respiratory syncytial virus (RSV), parainfluenza virus (PiV), human metapneumovirus (hMPV), and rhinovirus
* At least 6 months post-transplant, with completion of 6 month bronchoscopy if indicated
* Able and willing to give written informed consent and comply with study procedures (e.g. testing, treatment)

Exclusion Criteria:

* BOS Stage 3
* Requirement for mechanical ventilation at study entry
* Use of inhaled steroids at the time of CARV infection
* Any condition that in the investigator's opinion would preclude the patient's participation in a clinical trial
* Lack of available spirometric data to establish a baseline forced expiratory volume in 1 second and/or forced vital capacity
* Pregnancy
* Current participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramsey Hachem, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Beclomethasone | Placebo
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Beclomethasone | Placebo | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (20.7) | 62 (6.6) | 57.1 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Bronchiolitis Obliterans Syndrome Stage [Number; unit: participants]
  BOS Stage 0 or 0p (Forced expiratory volume in 1 second is at least 81% of baseline) | 7 | 6 | 13
  BOS Stage 1 or 2 (Forced expiratory volume in 1 second is between 51-80% of baseline) | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From New or Progressive Chronic Lung Allograft Dysfunction
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Beclomethasone | Placebo
Number analyzed (Participants) | 7 | 8
Participants | 2 | 4

2. Primary Outcome: Death
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Beclomethasone | Placebo
Number analyzed (Participants) | 7 | 8
Participants | 0 | 0

3. Secondary Outcome: Acute Rejection
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Beclomethasone | Placebo
Number analyzed (Participants) | 7 | 8
Participants | 1 | 0

4. Secondary Outcome: Lymphocytic Bronchiolitis
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Beclomethasone | Placebo
Number analyzed (Participants) | 7 | 8
Participants | 0 | 1

5. Secondary Outcome: Donor-specific Antibodies
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Beclomethasone | Placebo
Number analyzed (Participants) | 7 | 8
Participants | 0 | 0

6. Secondary Outcome: Chronic Lung Allograft Dysfunction
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Beclomethasone | Placebo
Number analyzed (Participants) | 7 | 7
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Inhaled Beclomethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/7 | 5/8
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Beclomethasone (N=7) | Placebo (N=8)
Chronic Lung Allograft Dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
New Respiratory Viral Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Lower Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Beclomethasone (N=7) | Placebo (N=8)
New Respiratory Viral Infection (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cold Symptoms (General disorders) | 1 (1) | 4 (4)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hoarseness (General disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin Cancer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Chronic Lung Allograft Dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Mycobacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT02351180/Prot_SAP_000.pdf